CLINICAL TRIAL: NCT03286088
Title: Mitral Valve Regurgitation Quantification From 3D Color Doppler Ultrasound - Standard of Care Data Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICBE-2-15217
Record Dates: First submitted 2017-03-31; First posted 2017-09-18 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Mitral Valve Regurgitation of Any Grade
MeSH Terms: interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Other): TransEsophageal Echocardiography + TransThoracic Echocardiography
  Interventions: Diagnostic Test: TransEsophageal Echocardiography and TransEsophageal Echocardiography
- Group B (Other): TransEsophageal Echocardiography + TransThoracic Echocardiography + cardiac Magnetic Resonance
  Interventions: Diagnostic Test: TransEsophageal Echocardiography and TransEsophageal Echocardiography; Diagnostic Test: Cardiac Magnetics Resonance
- Group C (Other): TransEsophageal Echocardiography + TransThoracic Echocardiography + MitraClip
  Interventions: Diagnostic Test: TransEsophageal Echocardiography and TransEsophageal Echocardiography; Diagnostic Test: MitraClip

INTERVENTIONS:
Diagnostic Test: TransEsophageal Echocardiography and TransEsophageal Echocardiography — imaging as standard practice
Diagnostic Test: Cardiac Magnetics Resonance — imaging as standard practice
  Arms: Group B
Diagnostic Test: MitraClip — imaging as standard practice
  Arms: Group C

SUMMARY:
The study primarily aims to collect standard of care clinical data in a wide spectrum of simple to complex mitral valve regurgitation (MVR) cases to validate a post-processing stand-alone software prototype (QFlow), developed by Philips Research Paris (Medisys).

Investigator does not intervene in the care of the patient, but simply collects standard of care images and measurements that are needed for the validation of the investigational software.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* age between 18 and 85 years old (adult, senior)
* sinus rhythm
* hHemodynamic stable
* mitral valve regurgitation (MVR) of any grade i.e., from mild to severe as determined by assessment of a qualifying TransThoracic Echocardiography (TTE) exam at Saint-Luc University Hospital
* scheduled for TransEsophageal Echocardiography (TEE) at Saint-Luc University Hospital, as part of the subject's routine standard of care
* subjects has functional capacity to give written informed consent

Exclusion Criteria:

* pregnancy
* subject lacks functional capacity to give written informed consent belongs to a vulnerable population per investigator's judgment or subject has any kind of disorder that compromises his/her ability to give written informed consent and/or to comply with study procedures

Among the120 subjects, there will be three (3) sub-groups as follows:

* a first sub-group (A) of 50 subjects with all inclusion criteria and none of the exclusion criteria
* a second sub-group (B) of 50 subjects with additional inclusion criterion: scheduled for cardiac Magnetic Resonance (cMR), as part of the subject's routine standard of care
* a third sub-group (C) of 20 subjects with additional inclusion criterion: scheduled for MitraClip transcatheter mitral valve repair (MitraClip) procedure as part of the subject's routine standard of care

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Central diastolic and systolic blood pressures | Day 1
  images and measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luc University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No